CLINICAL TRIAL: NCT00378391
Title: European Registry on Patients With ST-Elevation MI Transferred for Mechanical Reperfusion (PCI)With a Special Focus on Upstream Use of Abciximab
Brief Title: European Registry on STEMI Patients Transferred for PCI With Upstream Use of Abciximab - EuroTransfer Registry
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Foundation for Medical Research in Krakow, Poland (Unknown)
Other Study IDs: H4S-PL-O067
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2007-06-20 (Estimated); Status verified 2007-06

CONDITIONS: ST-Elevation Myocardial Infarction; Acute Coronary Syndrome
Keywords: ST-Elevation Myocardial Infarction; upstream abciximab; guideline adherence; hospital networking
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
EUROTRANSFER Registry is a prospective, international, web-based European Registry on Patients with ST-Elevation MI Transferred for Mechanical Reperfusion (PCI) with a Special Focus on Upstream Use of Abciximab.

This registry is designed to collect data on approximately 1800 patients during a 12 month enrollment period in up to 20 interventional cardiology centres with hospital transfer networks from all over Europe.

Analysis of this registry should allow to monitor transfer timelines of patients arriving to the cath-lab from the regional hospital with or without upstream start of abciximab and scheduled for mechanical reperfusion (PCI) as well as to monitor regional differences across Europe in regard to the impact that time of various stages of the treatment chain may have on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS:

* All consecutive STEMI patients >=18years arriving to the Cath Lab hospital (invasive facility center) from transfer.

  * Transfer with respect to this registry is defined as patients that reach the Cath Lab hospital:

    1. transferred from a surrounding regional community hospitals that the Cath Lab hospital has an established referral pattern with or
    2. after being picked-up by an ambulance which is equipped/staffed to provide specific medical therapy (like prehospital thrombolysis or upstream abciximab). Usually these have a physician or specifically trained nurse on board.

       CENTRES:
  * Provide 24 hour/7 days on duty PCI service.
  * Has an established regional hospital referral network with >=8 patients/month arriving from transfer (as defined above).
  * A rate of >=10% of these transfer patients who receive upstream abciximab before or during transfer to the Cath Lab hospital. Start of abciximab in the ER or CCU of the Cath Lab hospital will not be considered as upstream start of abciximab.

Exclusion Criteria:

* Patients who arrive to the Cath Lab from other pathways than those specified above (a. and b.), e.g. those who come by ambulances that do not provide specific medical therapy or arrive directly to the ER of the Cath Lab hospital by own feet/car will not be included in this registry.
* Patients from controlled clinical trials shall be included as long as their actual treatment is fully known. Thus, participants from randomized trials with blinded treatment cannot be included in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800
Dates: Start 2005-11; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, Assoc. Prof., Principal Investigator — Cardiac Catheterization Laboratories, Jagiellonian University Medical College; Zbigniew Siudak, MD, Study Chair — Cardiac Catheterization Laboratories, Jagiellonian University Medical College; Lukasz Partyka, MD, PhD, Study Director — KCRI
Locations (15):
- Helsinki University Central Hospital, Helsinki, Finland
- Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen, Germany
- Italy (5):
  - San Donato Hospital, Arezzo
  - Ospedale Carlo Poma, Mantova
  - Ospedale G.Pasquinucci, Massa
  - Santa Maria Nuova Hospital Reggio Emilia, Reggio Emilia
  - Ospedale S.Maria di Ca Foncello, Treviso
- Poland (4):
  - Cardiac Catheterization Laboratories Jagiellonian University Medical College, University Hospital, Krakow
  - Department of Interventional Cardiology, John Paul II Hospital, Krakow
  - Szpital Wojewodzki w Przemyslu, Przemyśl
  - Szpital im. Szczeklika Tarnow, Tarnów
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Clinico Universitario, Santiago de Compostela
- Linköping University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Dziewierz A, Siudak Z, Rakowski T, Kleczynski P, Zasada W, Dubiel JS, Dudek D. Impact of direct stenting on outcome of patients with ST-elevation myocardial infarction transferred for primary percutaneous coronary intervention (from the EUROTRANSFER registry). Catheter Cardiovasc Interv. 2014 Nov 15;84(6):925-31. doi: 10.1002/ccd.25266. Epub 2014 Jul 29. PMID 24155092
- [Derived] Dziewierz A, Siudak Z, Rakowski T, Kleczynski P, Dubiel JS, Dudek D. Early administration of abciximab reduces mortality in female patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention (from the EUROTRANSFER Registry). J Thromb Thrombolysis. 2013 Oct;36(3):240-6. doi: 10.1007/s11239-012-0826-3. PMID 23065325
- [Derived] Dziewierz A, Mielecki W, Siudak Z, Rakowski T, Janzon M, Birkemeyer R, Zasada W, Dubiel JS, Dudek D. Early abciximab administration before primary percutaneous coronary intervention improves clinical outcome in diabetic patients with ST-segment elevation myocardial infarction (EUROTRANSFER Registry). Atherosclerosis. 2012 Jul;223(1):212-8. doi: 10.1016/j.atherosclerosis.2012.04.018. Epub 2012 May 15. PMID 22658254
- [Derived] Siudak Z, Zawislak B, Dziewierz A, Rakowski T, Jakala J, Bartus S, Noworolnik B, Zasada W, Dubiel JS, Dudek D. Transradial approach in patients with ST-elevation myocardial infarction treated with abciximab results in fewer bleeding complications: data from EUROTRANSFER registry. Coron Artery Dis. 2010 Aug;21(5):292-7. doi: 10.1097/MCA.0b013e32833aa6d1. PMID 20453640
- [Derived] Dudek D, Siudak Z, Janzon M, Birkemeyer R, Aldama-Lopez G, Lettieri C, Janus B, Wisniewski A, Berti S, Olivari Z, Rakowski T, Partyka L, Goedicke J, Zmudka K; EUROTRANSFER Registry Investigators. European registry on patients with ST-elevation myocardial infarction transferred for mechanical reperfusion with a special focus on early administration of abciximab -- EUROTRANSFER Registry. Am Heart J. 2008 Dec;156(6):1147-54. doi: 10.1016/j.ahj.2008.08.004. Epub 2008 Oct 19. PMID 19033011